CLINICAL TRIAL: NCT06278519
Title: Cardiac MRI and Biological Samples at the Acute Phase of a Myocardial Infarction
Brief Title: CARdiAc Mri and BiOLogical samplEs at the Acute Phase of a Myocardial Infarction (CARAMBOLE)
Acronym: CARAMBOLE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Collaborators: Fédération Française de Cardiologie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CARAMBOLE
Record Dates: First submitted 2023-12-19; First posted 2024-02-26 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Myocardial Infarction
Keywords: cardiology
MeSH Terms: conditions — Myocardial Infarction | interventions — Blood Specimen Collection; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Blood and urinary collection, cardiac MRI (Experimental): Blood and urinary collection, cardiac MRI at inclusion during acute phase of STEMI, and one year after inclusion visit.
  Interventions: Biological: Blood, urinary and feces collection; Device: Cardiac MRI; Other: Quality of life and cognitive status questionnaire

INTERVENTIONS:
Biological: Blood, urinary and feces collection — Blood, urinary and feces collection, at inclusion during acute phase of STEMI, and one year after inclusion visit.
Device: Cardiac MRI — Cardiac MRI at the acute phase of STEMI (Day 5 +/- 3) and at 1-year follow-up
Other: Quality of life and cognitive status questionnaire — Quality of life and cognitive status questionnaire at the acute phase of STEMI and at 1-year follow-up

SUMMARY:
ST-Segment Elevation Myocardial infarction (STEMI) corresponding to acute occlusion of cornary artery is the most severe ischemic myocardial disease and a leading cause of mortality of heart failure worldwide. Although acute mortality from STEMI has decreased over the last decades, the prognosis remains pejorative and difficult to anticipate. The best management of STEMI patients depends of predictive factors of clinical prognosis and justifies an active research of these factors, in particular the mechanisms leading to deleterious left ventricular remodeling, myocardial inflammation, reperfusion injury including the no-reflow phenomenon which is a major determinant of heart failure. Cohorts of consecutive STEMI patients, with a comprehensive assessment of clinical, biological and imaging parameters are needed to offer the basis for new hypothese for research or interventions and to precisely evaluate the quality of care provided.

The main objective of this study is to identify new markers: clinical, biological and imaging, treatment response and prognosis after STEMI.

Secondary objectives of the CARAMBOLE cohort are to establish a comprehensive clinical databse, completed with biological samples and imaging data, that can be used in the following areas:

* Descriptive epidemiology of STEMI and myocardial reperfusion
* Evaluation of the clinical implications of the realization of a cardiac MRI at the acute phase of STEMI (regarding no-reflow, LVEF, intra cardiac thrombi)
* Treatments observatory: safety, efficacy, indication of treatments provided in real life compared to the treatments recommended, adherence to treatments, costs
* Quality of life, personal, familial, social and professional consequences of myocardial infarction
* Research of new diagnostic and prognosis biomarkers
* Research projects (e.g risk of developping cgnitive disorders in patients with STEMI as compared to the general population)

Participants will undergo:

* a cardiac MRI at the acute phase of their STEMI (5 +/- 3 days) then at 1 year follow-up
* biological samples including blood, urinary and feces samples, at the acute phase of their STEMI (from admission and up to 8 days) then at 1 year follow-up
* questionnaire assessment regarding their quality of life, cognitive status,and socio-economic conditions at the acute phase and 1 year follow-up of their STEMI.

DETAILED DESCRIPTION:
Myocardial infarction is one of the leading causes of morbi-mortality, causing 75% of cases of sudden death in adults over 35 years of age and more than half of chronic heart failure. Despite the progress made, based on French data from the CIRCUS study and the FAST-MI registry, all-cause mortality at 1 year remained high at around 8% and the rate of occurrence of composite events (death, heart failure, myocardial infarction, revascularization, stroke) estimated around 25%. ST-segment elevation myocardial infarction (STEMI) is the most severe form of ischemic myocardial disease. The recommended treatment is the quickest possible unblocking of the coronary artery responsible for STEMI, by coronary angioplasty (treatment of choice if time limits are compatible) or, more rarely, thrombolysis. However, this revascularization causes undesirable collateral effects with tissue edema, intra-myocardial hemorrhages, microvascular obstruction and local inflammation which contribute to significantly aggravate myocardial damage. These "reperfusion injuries" increase the risk of Left Ventricular (LV) dysfunction. Thus, immediate mortality decreases but the incidence of heart failure following STEMI increases. Several other parameters associated with a poor prognosis remain to this day incompletely understood and treated: deleterious left ventricular remodeling (LVR), post-infarction inflammation, no-reflow.

Furthermore, performing a systematic MRI at the acute phase of STEMI will allow to assess the real prevalence of intra LV thrombi and to treat them before hospital discharge. Indeed, the prevalence of intraLV thrombi is estimated around 20% but only 16% are diagnosed during the stay in the Cardiology Intensive Care Unit (CICU) (low sensitivity of echocardiography, lack of availability of cardiac MRI) . These patients must be treated with anticoagulants to limit the embolic phenomena of intra LV thrombi, in particular strokes, but most patients therefore do not benefit from this treatment when leaving the hospital since MRI is not performed in the acute phase in most centers due to lack of availability.

The organization of prospective cohorts with well-documented biological and imaging collections, in particular the systematic use of myocardial MRI, and monitoring of events at 1 year, will thus make it possible to better understand the complex pathophysiology of these deleterious phenomena, their clinical consequences, to propose research hypotheses and ultimately, to developp innovative and personalized treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥18 years old, hospitalised in cardiology departments at the C.H.U. of Poitiers
* Myocardial infarction type 1, 2 or 3 according to the 4th universal definition, with elevation of ST segment ≥0.2 milliVolt in two contiguous derivations of the ECG.
* Patient able to comply with study procedures
* Patient legally free and not subject to any custody, guardianship, tutelage or subordination measures
* Informed consent signed by the patient/relative or trusted person after clear and complete information about the clinical investigation.

Exclusion Criteria:

* Subject with contraindication to MRI : pregnancy, ocular metallic foreign body (accidental or other chips), pace-maker incompatible with MRI, foreign ferromagnetic ocular or cerebral bodies, cochlear implants and in general all electronic medical material immovably implanted and incompatible with MRI; metallic heart valve of 1st generation, vascular clips formerly implanted on cranial aneurysm, severe renal insufficiency
* Patient suffering from claustrophobia
* Hypersensitivity to gadoteric acid, to meglumine or to a drug containing gadolinium
* patients with insufficient venous access for contrast medium injection.
* Participation in another interventional study with an investigational drug or device, which, in the judgment of the investigator, could interfere with the present study
* Patients not benefiting from a Social Security scheme or not benefiting from it through a third party
* Persons benefitting from enhanced protection, namely minors, pregnant women, persons deprived of their liberty by a judicial or administrative decision, patients staying in a health or social establishment, adults under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Major Adverse cardiac Events (MACE) | Up to 1 year after STEMI
  MACE (death, recurrence of myocardial infarction, ischemic stroke, hospitalization for heart failure, unplanned coronary revascularization) will be assessed through medical records and clinical follow-up

SECONDARY OUTCOMES:
Infarct size | Up to 8 days after STEMI
  Infarct size will be measured on Cardiac MRI
Infarct size | 1 year follow-up after STEMI
  Infarct size will be measured on Cardiac MRI
No-reflow size | Up to 8 days after STEMI
  No-reflow size will be measured on Cardiac MRI
No-reflow size | 1 year follow-up after STEMI
  No-reflow size will be measured on Cardiac MRI
Cardiac enzymes rate | H0 (admission in Intensive Cardiac Care Unit)
  Cardiac enzymes rate will be analyzed on blood samples
Cardiac enzymes rate | H24 (24 hours after reperfusion)
  Cardiac enzymes rate will be analyzed on blood samples
Cardiac enzymes rate | H48 (48 hours after reperfusion)
  Cardiac enzymes rate will be analyzed on blood samples
Cardiac enzymes rate | 1 year follow-up after STEMI
  Cardiac enzymes rate will be analyzed on blood samples
Inflammatory markers rate | H0 (admission in Intensive Cardiac Care Unit)
  Inflammatory markers rate will be analyzed on blood samples
Inflammatory markers rate | H24 (24 hours after reperfusion)
  Inflammatory markers rate will be analyzed on blood samples
Inflammatory markers rate | H48 (48 hours after reperfusion)
  Inflammatory markers rate will be analyzed on blood samples
Inflammatory markers rate | 1 year follow-up after STEMI
  Inflammatory markers rate will be analyzed on blood samples
Gut microbiota profiling | Up to 8 days after STEMI
  Gut microbiota will be assessed on feces samples. Metagenomic sequencing and 16S ribosomal ribonuleic acid (RNA) gene sequencing will be applied to investigate gut microbiota richness, diversity and composition.
Gut microbiota profiling | 1 year follow-up after STEMI
  Gut microbiota will be assessed on feces samples. Metagenomic sequencing and 16S ribosomal ribonuleic acid (RNA) gene sequencing will be applied to investigate gut microbiota richness, diversity and composition.
Genitourinary microbiota profiling | Up to 8 days after STEMI
  Genitourinary microbiota will be assessed on urine samples. Metagenomic sequencing and 16S ribosomal ribonuleic acid (RNA) gene sequencing will be applied to investigate genitourinary microbiota richness, diversity and composition.
Genitourinary microbiota profiling | 1 year follow-up after STEMI
  Genitourinary microbiota will be assessed on feces samples. Metagenomic sequencing and 16S ribosomal ribonuleic acid (RNA) gene sequencing will be applied to investigate genitourinary microbiota richness, diversity and composition.
EQ-5D-3L score (European Quality of Life 5 Dimensions 3 Level version) | Up to 8 days after STEMI
  Patients' quality of life will be evaluated by the EQ-5D-3L questionnaire, which ranges from 5 to 15, with a highest score meaning a worse outcome
EQ-5D-3L score (European Quality of Life 5 Dimensions 3 Level version) | 1 year follow-up after STEMI
  Patients' quality of life will be evaluated by the EQ-5D-3L questionnaire, which ranges from 5 to 15, with a highest score meaning a worse outcome
Codex test | Up to 8 days after STEMI
  Patients' cognitive status will be evaluated by the Codex test
Codex test | 1 year follow-up after STEMI
  Patients' cognitive status will be evaluated by the Codex test

CONTACTS AND LOCATIONS:
Locations (1):
- C.H.U. of Poitiers, Poitiers, France